CLINICAL TRIAL: NCT03601793
Title: Using Assistance From a Health Educator to Increase Effectiveness of an Internet Intervention for Alcohol Problems. A Randomized Controlled Trial
Brief Title: An Internet Intervention for Alcohol Problems With or Without Assistance From a Health Educator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 029/2018
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Alcohol Problem
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet intervention with assistance (Experimental): This arm is given access to the internet intervention Alcohol Help Center with email assistance from a health educator during the first two weeks after randomization.
  Interventions: Behavioral: Alcohol Help Center; Behavioral: Assistance from a health educator
- Internet intervention without assistance (Active Comparator): This arm is given access to the internet intervention Alcohol Help Center without any assistance from a health educator.
  Interventions: Behavioral: Alcohol Help Center

INTERVENTIONS:
Behavioral: Alcohol Help Center — An internet intervention based on CBT consisting of about 20 modules aimed at helping people with drinking problems
Behavioral: Assistance from a health educator — This entails email contact with a health educator that guides the participant through the Alcohol Help Center during the first two weeks
  Arms: Internet intervention with assistance

SUMMARY:
The purpose of this study is to determine whether an internet intervention for alcohol problems is more effective when delivered with assistance from a health care educator via e-mail during the first two weeks after randomization, as compared to simply providing the intervention without any such assistance.

DETAILED DESCRIPTION:
This project aims to study the previously evaluated multi-module internet intervention Alcohol Help Center delivered with assistance from a health educator (AHC+A). The assistance will be in the form of email contact with the participant during the first two weeks after randomization. AHC+A will be tested against a group receiving access to the intervention without any such assistance (AHC).

The Investigators hypothesize that

1. participants allocated to AHC+A will display significant reductions in drinking (drinks preceding week/heavy drinking days preceding week) in 3- and 6-month follow ups compared to AHC
2. participants allocated to AHC+A will display greater engagement with the intervention in terms of a higher number of modules completed compared to AHC
3. engagement with the intervention will mediate any effects on drinking behavior.

A 2-arm parallel group randomized controlled trial will be used to test these specified hypotheses. Follow-ups will be conducted at 3 and 6 months after randomization. Online media advertisements will be used to recruit people with current alcohol problems, and will target people who are 'experiencing difficulties in controlling or cutting down on their drinking.' The advertisements will be placed across Canada using locations found successful in previous trials to rapidly recruit participants (e.g. Google AdWords).

ELIGIBILITY:
Inclusion Criteria:

* A score of 8 or more on the Alcohol Use Disorder Identification Test (AUDIT)
* A preceding week alcohol consumption of 14 standard drinks or more

Exclusion Criteria:

* Being under 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Drinks preceding week | 3 and 6 months
  Change in the number of standard drinks consumed during preceding week from baseline
Heavy drinking days preceding week | 3 and 6 months
  Change in the number of heavy drinking days during preceding week from baseline

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline, 3 month follow up, 6 month follow up
  Assessment of alcohol problems
Alcohol Use Disorders Identification Test - Consumption (AUDIT-C) | Baseline, 3 month follow up, 6 month follow up
  Assessment of alcohol consumption (the first 3 items in AUDIT)
EuroQol Group 5 Dimensions Five Levels (EQ-5D-5L) | Baseline, 3 month follow up, 6 month follow up
  Instrument measuring five health-related quality of life dimensions. Each dimension has five levels ranging from no problems to extreme problems. The dimensions can be combined into an index value between 0 (lowest) and 1 (highest). In addition to the five dimensions, a visual analogue scale item allows participants to measure health outcomes that reflect the participant's judgement. Endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
DSM criteria | Baseline
  The 11 DSM criteria of alcohol use disorders (yes/no)
Previously received treatment or help for alcohol concerns | Baseline (treatment or help ever/in the past 12 months), 3 month follow up (treatment or help in the past 3 months), 6 month follow up (treatment or help in the past 3 months)
  Questions about what kind of treatment or help for alcohol concerns the participant has received previously

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research